CLINICAL TRIAL: NCT00440297
Title: A Study in Renal Predialysis and Dialysis Patients of the Safety, Tolerability, and Immunogenicity of Recombinant Hepatitis B Vaccine Manufactured With a Modified Process
Brief Title: Hepatitis B Vaccine Predialysis/Dialysis Study (V232-060)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V232-060; 2007_515 (Other: Merck Registration Number)
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Results first posted 2009-07-08 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B Virus Infection
Keywords: hepatitis B virus
MeSH Terms: conditions — Hepatitis B

ARMS (2):
- Modified process hepatitis B vaccine (Experimental): Modified process hepatitis B vaccine 40 ug/1.0 mL injection in a 4 dose regimen at months 0, 1, 6, and 8. Duration of treatment is 9 months.
  Interventions: Biological: Comparator: modified process hepatitis B vaccine
- ENGERIX-B™2 (Active Comparator): ENGERIX-B™ two 20 ug/1.0 mL injections in a 4 dose regimen at months 0, 1, 6, and 8. Duration of treatment is 9 months.
  Interventions: Biological: Comparator: ENGERIX-B™

INTERVENTIONS:
Biological: Comparator: modified process hepatitis B vaccine — Modified process hepatitis B vaccine 40 ug/1.0 mL injection in a 4 dose regimen at months 0, 1, 6, and 8. Duration of treatment is 9 months.
  Arms: Modified process hepatitis B vaccine
Biological: Comparator: ENGERIX-B™ — ENGERIX-B™ two 20 ug/1.0 mL injections in a 4 dose regimen at months 0, 1, 6, and 8. Duration of treatment is 9 months.
  Arms: ENGERIX-B™2

SUMMARY:
To describe the immunogenicity and safety of modified process hepatitis B vaccine administered to renal predialysis and dialysis patients

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects at least 18 years of age
* Laboratory confirmed negative serology result to HbsAg (hepatitis b virus), anti-HBs (antibody to hepatitis B surface antigen), and anti HBc (antibody to hepatitis B core antigen) within 6 weeks of the initial dose of study vaccine
* Patient on renal dialysis or a pre-dialysis patient with a creatinine clearance of <=30 ml/min

Exclusion Criteria:

* Previous hepatitis B infection, vaccination with any hepatitis B vaccine
* Recent febrile illness; hypersensitivity to any component of licensed hepatitis B vaccines
* Recent administration of immune globulin, licensed inactivated vaccine within 14 days or licensed live vaccine within 30 days prior to receipt of first study vaccine
* Receipt of investigational drugs or investigational vaccines within 3 months prior
* Impairment of immunologic function
* Recent use of systemic immunomodulatory medications
* Pregnant women, nursing mothers or women planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2006-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Gilbert CL, Stek JE, Villa G, Klopfer SO, Martin JC, Schodel FP, Bhuyan PK. Safety and immunogenicity of a recombinant hepatitis B vaccine manufactured by a modified process in renal pre-dialysis and dialysis patients. Vaccine. 2014 Nov 12;32(48):6521-6. doi: 10.1016/j.vaccine.2014.09.015. Epub 2014 Sep 22. PMID 25252192

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22-Dec-2006 (First Patient Enrolled in Study) to 05-May-2008 (Last Participant had their Last Visit). This study was conducted at 23 sites: 7 in Canada, 8 in the United Kingdom, 5 in Italy, and 3 in Spain. In the Modified Process group, one participant was randomized by mistake, and therefore was not vaccinated.
Pre-assignment Details: A screening serum sample was obtained prior to study entry and assayed for hepatitis B serologic markers. Only patients that were seronegative were considered for enrollment.
Groups:
- Modified Process Hepatitis B Vaccine: Modified Process Hepatitis B Vaccine, 40 µg(micrograms)
- ENGERIX-B™: ENGERIX-B™, 2 x 20 µg(micrograms)
Period: Overall Study
Arm/Group | Modified Process Hepatitis B Vaccine | ENGERIX-B™
Started | 139 | 138
Vaccination Visit 1 | 138 | 138
Vaccination Visit 2 | 136 | 134
Vaccination Visit 3 | 124 | 125
Vaccination Visit 4 | 116 | 122
Completed | 116 | 120
Not Completed | 23 | 18
Not completed — Adverse Event | 8 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 11 | 7
Not completed — Withdrawal by Subject | 1 | 6
Not completed — Randomized by mistake | 1 | 0

BASELINE CHARACTERISTICS:
Population: All vaccinated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Process Hepatitis B Vaccine | ENGERIX-B™ | Total
Number analyzed (Participants) | 138 | 138 | 276
Age, Continuous [Mean (Full Range); unit: years] | 69.7 [20 to 91] | 69.2 [30 to 90] | 69.5 [20 to 91]
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.7 (13.4) | 69.2 (12.7) | 69.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 56 | 109
  Male | 85 | 82 | 167

OUTCOME MEASURES:

1. Primary Outcome: The Number of Seroprotected Participants to the Modified Process Hepatitis B Vaccine and ENGERIX-B™ (Currently Licensed Vaccine) at Month 7
Description: The number of participants as measured by the
  seroprotection rate (anti-hepatitis B surface antibodies greater than or equal to 10 mIU/mL). Anti-HBs (Antibodies against hepatitis B surface antigen) titers were measured from blood samples taken at Day 1 (prior to the first dose) and at Month 7 (1 month after the third dose).
Time Frame: 7 months (1 month after the third dose)
Population: Per-Protocol Population: The Per-Protocol Population is defined as the participants that were able to complete the study as defined by the protocol.
Measure: Number; unit: Participants
Arm/Group | Modified Process Hepatitis B Vaccine | ENGERIX-B™
Number analyzed (Participants) | 101 | 111
Participants | 49 | 64
Statistical Analysis 1: Comparison: Modified Process Hepatitis B Vaccine; No hypothesis is being tested. The purpose of the primary analysis is to estimate the seroprotection rate (percentage of subjects with anti-HBs >=10mIU/mL) in each group at 1 month after the third dose among subjects who were seronegative at baseline; Test type: Superiority or Other; Percentage of Seroprotected Participants = 48.5, 95% CI [38.4 to 58.7] — Exact binomial confidence interval
Statistical Analysis 2: Comparison: ENGERIX-B™; Test type: Superiority or Other; Percentage of Seroprotected Participants = 57.7, 95% CI [47.9 to 67.0] — Exact binomial confidence interval

2. Primary Outcome: The Number of Seroprotected Participants to the Modified Process Hepatitis B Vaccine and ENGERIX-B™ (Currently Licensed Vaccine) at Month 9
Description: The number of participants as measured by the
  seroprotection rate (anti-hepatitis B surface antibodies greater than or equal to 10 mIU/mL). Anti-HBs (Antibodies against hepatitis B surface antigen) titers were measured from blood samples taken at Day 1 (prior to the first dose) and at Month 9 (1 month after the fourth dose).
Time Frame: 9 months (1 month after the fourth dose)
Population: Per-Protocol Population: The Per-
  Protocol Population is defined as the participants that were able to complete the study as defined by the
  protocol.
Measure: Number; unit: Participants
Arm/Group | Modified Process Hepatitis B Vaccine | ENGERIX-B™
Number analyzed (Participants) | 99 | 104
Participants | 66 | 72
Statistical Analysis 1: Comparison: Modified Process Hepatitis B Vaccine; Test type: Superiority or Other; Percentage of Seroprotected Participants = 66.7, 95% CI [56.5 to 75.8] — Exact binomial confidence interval
Statistical Analysis 2: Comparison: ENGERIX-B™; Test type: Superiority or Other; Percentage of Seroprotected Participants = 69.2, 95% CI [59.4 to 77.9] — Exact binomial confidence interval

3. Primary Outcome: The Total Number of Participants With One or More Injection-Site Adverse Experiences
Time Frame: Days 1-15 After Any Vaccination
Population: Safety Analysis Set: The Safety Analysis Set is defined as all participants who receive at least one injection of vaccine and who had a safety follow-up
Measure: Number; unit: Participants
Arm/Group | Modified Process Hepatitis B Vaccine | ENGERIX-B™
Number analyzed (Participants) | 138 | 135
Participants | 43 | 48

4. Primary Outcome: The Total Number of Participants With a Maximum Temperature >= 100.0F / 37.8C
Time Frame: Days 1-5 After Any Vaccination
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Modified Process Hepatitis B Vaccine | ENGERIX-B™
Number analyzed (Participants) | 138 | 135
Participants | 5 | 6

5. Primary Outcome: The Total Number of Participants With Serious Vaccine-Related Clinical Adverse Experiences
Description: Participants with adverse experiences considered possibly, probably, or definitely related to study vaccines and considered serious (death, persistent disability, life threatening, hospitalization, birth defects, cancer, or overdose).
Time Frame: 0-9 months (recorded from first dose until the participant completes or discontinues the study)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Modified Process Hepatitis B Vaccine | ENGERIX-B™
Number analyzed (Participants) | 138 | 135
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events: Days 1-15 after any vaccination; Deaths and vaccine-related serious adverse events: up to 9 months
Arm/Group | Modified Process Hepatitis B Vaccine | ENGERIX-B™
Serious Adverse Events (participants affected / at risk) | 11 | 11
Other Adverse Events (participants affected / at risk) | 56 | 73
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Modified Process Hepatitis B Vaccine | ENGERIX-B™
Pneumonia (Infections and infestations) | 2/138 | 0/135
Myocardial Infarction (Cardiac disorders) | 4/138 | 2/135
Hip fracture (Injury, poisoning and procedural complications) | 1/138 | 0/135
Anaemia (Blood and lymphatic system disorders) | 1/138 | 1/135
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1/138 | 0/135
Cerebral ischaemia (Nervous system disorders) | 1/138 | 0/135
Renal failure (Renal and urinary disorders) | 1/138 | 2/135
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/138 | 0/135
Pancreatitis acute (Gastrointestinal disorders) | 1/138 | 0/135
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1/138 | 0/135
Hepatitis (Hepatobiliary disorders) | 1/138 | 0/135
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1/138 | 0/135
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/138 | 0/135
Liver function test abnormal (General disorders) | 1/138 | 0/135
Cardiac failure congestive (Cardiac disorders) | 0/138 | 1/135
Cardiac arrest (Cardiac disorders) | 0/138 | 1/135
Gastric ulcer (Gastrointestinal disorders) | 0/138 | 1/135
Cardio-respiratory arrest (Cardiac disorders) | 0/138 | 1/135
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0/138 | 1/135
Renal failure chronic (Renal and urinary disorders) | 0/138 | 1/135
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0/138 | 1/135
Renal haematoma (Injury, poisoning and procedural complications) | 0/138 | 1/135
Circulatory collapse (Vascular disorders) | 0/138 | 1/135
Sepsis (Infections and infestations) | 0/138 | 2/135
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0/138 | 1/135
Hypoglycaemia (Metabolism and nutrition disorders) | 0/138 | 1/135
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Modified Process Hepatitis B Vaccine | ENGERIX-B™
Constipation (Gastrointestinal disorders) | 2/138 | 1/135
Diarrhea (Gastrointestinal disorders) | 5/138 | 6/135
Nausea (Gastrointestinal disorders) | 3/138 | 2/135
Vomiting (Gastrointestinal disorders) | 2/138 | 1/135
Asthenia (General disorders) | 1/138 | 2/135
Fatigue (General disorders) | 4/138 | 1/135
Edema peripheral (General disorders) | 1/138 | 3/135
Pyrexia (General disorders) | 4/138 | 6/135
Cystitis (Infections and infestations) | 2/138 | 0/135
Lower respiratory tract infection (Infections and infestations) | 0/138 | 2/135
Nasopharyngitis (Infections and infestations) | 2/138 | 3/135
Urinary tract infection (Infections and infestations) | 0/138 | 3/135
Athralgia (Musculoskeletal and connective tissue disorders) | 3/138 | 4/135
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2/138 | 1/135
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2/138 | 1/135
Dizziness (Nervous system disorders) | 4/138 | 5/135
Headache (Nervous system disorders) | 8/138 | 8/135
Insomnia (Psychiatric disorders) | 0/138 | 4/135
Cough (Respiratory, thoracic and mediastinal disorders) | 2/138 | 2/135
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2/138 | 0/135
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0/138 | 2/135
Pruritis (Skin and subcutaneous tissue disorders) | 1/138 | 2/135
Injection site Erythema (General disorders) | 7/138 | 19/135
Injection site Edema (General disorders) | 1/138 | 2/135
Injection site Pain (General disorders) | 32/138 | 39/135
Injection site Swelling (General disorders) | 12/138 | 14/135

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.